CLINICAL TRIAL: NCT02579811
Title: A Phase II Study of the Efficacy and Safety of Axitinib Given on an Individualized Schedule for Metastatic Renal Cell Cancer After Treatment With Pd-1 or Pd-L1 Inhibitors
Brief Title: Axitinib Given on an Individualized Schedule for Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE7815
Record Dates: First submitted 2015-10-14; First posted 2015-10-20 (Estimated); Results first posted 2020-08-07 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Metastatic Renal Cell Cancer
Keywords: Kidney; Cancer; Axitinib; Pd-1 inhibitor; Pd-L1 inhibitor
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Axitinib (Experimental): All subjects will be given axitinib on an individualized dosing schedule. Axitinib will be administered orally beginning with 5mg twice a day and can be escalated or reduced if specific grade 2 or greater toxicity develops. Axitinib will continue until progression. At progressive disease, dose escalation above current dose is allowed based on investigator discretion of clinical benefit. However, axitinib should be discontinued if a subject experiences a second RECIST progressive disease following dose escalation, patient intolerability, or at provider discretion.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — The intent is to maximize sustained dose intensity of axitinib based on individual tolerability using dose modification criteria

SUMMARY:
Axitinib is a drug which is approved by the FDA for patients with advanced kidney cancer who have already received some treatment. It works by reducing blood flow to a tumor. Axitinib is normally give at 5mg twice per day and sometimes this dose is increased if patients tolerate it. The purpose of this study is to figure out a different way to decide which dose of axitinib each patient should receive based on the side effects they experience.

DETAILED DESCRIPTION:
Primary objective To determine whether axitinib given on an individualized dose/schedule for metastatic renal cell carcinoma following immunotherapy with PD-1 and PD-L1 Inhibitors leads to improved progression-free survival (PFS).

Secondary objectives:

1. To characterize the objective response rates in patients given axitinib on an individualized dose/schedule.
2. To evaluate the tolerability and safety of an alternative method of axitinib titration.
3. To characterize the anti-tumor effect, as measured by change in tumor burden per RECIST 1.1, of axitinib titration performed after initial RECIST PD on axitinib.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, locally recurrent or metastatic clear cell renal cell carcinoma
* Has received one prior systemic therapy regimen for Metastatic Renal Cell Carcinoma (mRCC) directed against PD-1 and/or PD-L1 which must have been the most recent regimen

  * Prior high-dose interleukin-2 therapy is permitted in addition to anti-PD(L)1 therapy, but is not required
  * Prior bevacizumab or Vascular Endothelial Growth Factor (VEGF) Tyrosine Kinas Inhibitor (TKI) is permitted either in combination with anti-PD(L)1 therapy OR as monotherapy when given PRIOR to anti-PD(L)1 therapy
  * Prior treatment with combined ipilimumab and nivolumab is permitted
  * Prior axitinib in any setting is not permitted
  * A minimum of two weeks since last dose of most recent renal cell cancer therapy assuming resolution of clinically significant treatment-related toxicities to grade 1, baseline, or controlled with supportive medications
* Evidence of measurable disease per RECIST 1.1.
* Karnofsky performance status ≥ 70 %.
* Adequate organ function as defined by:

  * Absolute neutrophil count (ANC) ≥1,000/μL
  * Platelets ≥100,000/μL
  * Hemoglobin ≥9.0 g/dL
  * Serum calcium ≤12.0 mg/dL
  * Serum creatinine ≤2.0 x Upper Limit of Normal (ULN)
  * Total serum bilirubin ≤1.5 x ULN
  * SGOT≤2.5 x ULN and Serum Glutamic Pyruvic Transaminase (SGPT) ≤2.5x ULN
* Signed informed consent and willingness/ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

* Non clear cell Renal Cell Carcinoma (RCC)
* Major surgery within 4 weeks of starting the study treatment.
* Radiation therapy within 2 weeks of starting the study treatment. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been irradiated.
* NCI CTCAE Version 4.03 grade 3 hemorrhage within 4 weeks of starting the study treatment.
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack.
* Ongoing cardiac dysrhythmias of NCI CTCAE Version 4.03 grade ≥2. Controlled atrial fibrillation is permitted.
* Uncontrolled hypertension (>160/100 mm Hg despite optimal medical therapy)
* Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials, e.g. QOL, and imaging trials, are allowed.
* Pregnancy or breastfeeding. Female subjects must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the period of therapy. All female subjects with reproductive potential must have a negative pregnancy test (serum) prior to enrollment. Male subjects must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
* Uncontrolled Central Nervous System (CNS) metastases. Patients are considered to have controlled CNS metastases (and thus eligible) if they have completed local therapy (XRT and/or surgery) and are off steroids with clinical and radiographic stability 3 months from the end of CNS-directed therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12-30 (Actual); Primary Completion 2019-08-21 (Actual); Study Completion 2023-06-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Ornstein, MD, MA, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (4):
- United States (4):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio
  - The Ohio State University Comprehensive Cancer Center - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute, Columbus, Ohio
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] Ornstein MC, Pal SK, Wood LS, Tomer JM, Hobbs BP, Jia XS, Allman KD, Martin A, Olencki T, Davis NB, Gilligan TD, Mortazavi A, Rathmell WK, Garcia JA, Rini BI. Individualised axitinib regimen for patients with metastatic renal cell carcinoma after treatment with checkpoint inhibitors: a multicentre, single-arm, phase 2 study. Lancet Oncol. 2019 Oct;20(10):1386-1394. doi: 10.1016/S1470-2045(19)30513-3. Epub 2019 Aug 16. PMID 31427205

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Axitinib
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants who went on study
Arm/Group | Axitinib
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 23
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 6
  Male | 21
  Unknown | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 13
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Median Progression-free Survival
Description: The primary endpoint of progression-free survival in months (per per RECIST v1.1 criteria) will be estimated using the Kaplan-Meier method. Summary statistics will be provided along with 95% confidence intervals.
Time Frame: Up to 18 months
Population: Participants who went on study
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib
Number analyzed (Participants) | 40
months | 8.8 [5.7 to 16.6]

2. Secondary Outcome: Patients With Complete Response
Description: Tumor Response, defined as overall confirmed objective response, is confirmed complete response (CR) according to the RECIST 1.1 criteria. RECIST 1.1: Complete response (CR) is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Time Frame: Up to 4 months of treatment and approximately 1 year of follow-up
Population: Participants who went on study
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib
Number analyzed (Participants) | 40
Participants | 1

3. Secondary Outcome: Patients With Partial Response
Description: Tumor Response, defined as overall confirmed objective response, is confirmed complete response (CR) according to the RECIST 1.1 criteria. RECIST 1.1: Partial response (PR) is defined as a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Up to 4 months of treatment and approximately 1 year of follow-up
Population: Participants who went on study
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib
Number analyzed (Participants) | 40
Participants | 17

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR as defined by Recist V. 1.1. ORR = (CR + PR)
Time Frame: Up to 4 months of treatment and approximately 1 year of follow-up
Population: Participants who went on study
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib
Number analyzed (Participants) | 40
Participants | 18

ADVERSE EVENTS:
Time Frame: Up to 4 months of treatment and approximately 30 days of additional follow-up
Description: All serious adverse events collected and all adverse events related to the study drug.
Arm/Group | Axitinib
All-Cause Mortality (participants affected / at risk) | 13/40
Serious Adverse Events (participants affected / at risk) | 20/40
Other Adverse Events (participants affected / at risk) | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axitinib (N=40)
Dehydration (Metabolism and nutrition disorders) | 6 (10)
Diarrhea (Gastrointestinal disorders) | 3 (5)
Hypotension (Cardiac disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (2)
Hyperkalemia (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Bone infection (Infections and infestations) | 1 (2)
Fournier's gangrene (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (2)
Adrenal insufficiency (Endocrine disorders) | 1 (2)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (2)
Pain (General disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (2)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=40)
Fatigue (General disorders) | 33
Hypertension (Cardiac disorders) | 30
Hand-foot syndrome (Gastrointestinal disorders) | 26
Decreased appetite (Metabolism and nutrition disorders) | 24
Diarrhea (Gastrointestinal disorders) | 23
Dysphonia (General disorders) | 22
Nausea or vomiting (Gastrointestinal disorders) | 20
Constipation (Gastrointestinal disorders) | 19
Hypothyroidism (Endocrine disorders) | 17
Elevated creatinine (Blood and lymphatic system disorders) | 17
Arthralgia or myalgia (Musculoskeletal and connective tissue disorders) | 13
Anaemia (Blood and lymphatic system disorders) | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Mucositis (Gastrointestinal disorders) | 5
Elevated haemoglobin (Blood and lymphatic system disorders) | 4
Weight loss (General disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 2
Headache (General disorders) | 2
Elevated lipase (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT02579811/Prot_SAP_002.pdf
  • Informed Consent Form (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT02579811/ICF_001.pdf